CLINICAL TRIAL: NCT05629546
Title: Phase I Study of Memory-Like Natural Killer Cells With Nivolumab and Relatlimab in Advanced or Metastatic Melanoma After Progression on Checkpoint Inhibitors
Brief Title: Memory-Like Natural Killer Cells With Nivolumab and Relatlimab in Advanced or Metastatic Melanoma After Progression on Checkpoint Inhibitors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Melanoma Research Alliance (Other); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202404189
Record Dates: First submitted 2022-11-16; First posted 2022-11-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Melanoma; Metastatic Melanoma
Keywords: advanced melanoma; metastatic melanoma; checkpoint inhibitor resistant melanoma
MeSH Terms: conditions — Melanoma | interventions — Opdualag; Nivolumab

STUDY DESIGN:
Intervention Model Description: Enrollment will occur in parallel into arms 1 and 2, but sequence of enrollment will be staggered for the first 3 patients, with sequential patients being enrolled upon the previous patient completing 30 days of observation. Approximately 11 allogeneic donors will also be enrolled for subjects in Arm 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Autologous: Memory-like natural killer cells + nivolumab + relatilimab (Experimental): * Subjects enrolled into arm 1 will receive autologous ML NK cells on Day 0.
  * Relatlimab and nivolumab will be initiated at day 29 and continue every 28 days for 11 cycles, or until unacceptable toxicity, or progression, whichever is earlier.
  Interventions: Biological: Cytokine-induced memory-like natural killer cells; Biological: Relatilmab; Biological: Nivolumab
- Arm 2: Allogeneic: Memory-like natural killer cells + nivolumab + relatilimab (Experimental): * Subjects with a haploidentical donor will enroll into Arm 2
  * Subjects will receive the IV infusion of ML NK cells on Day 0.
  * Relatlimab and nivolumab will be initiated at day 29 and continue every 28 days for 11 cycles, or until unacceptable toxicity, or progression, whichever is earlier.
- Allogeneic Donors (No Intervention)

INTERVENTIONS:
Biological: Cytokine-induced memory-like natural killer cells — Cell product processing is performed at the Siteman Cancer Center Biological Therapy Core Facility (BTCF).
  Other Names: ML NK cells; CIML
  Arms: Arm 1: Autologous: Memory-like natural killer cells + nivolumab + relatilimab
Biological: Relatilmab — Standard of care
  Other Names: Opdualag
  Arms: Arm 1: Autologous: Memory-like natural killer cells + nivolumab + relatilimab
Biological: Nivolumab — Standard of care
  Arms: Arm 1: Autologous: Memory-like natural killer cells + nivolumab + relatilimab

SUMMARY:
This is a Phase 1 open-label, study designed to characterize the safety, tolerability, and preliminary anti-tumor activity of memory-like natural killer cells (ML NK) in combination with nivolumab and relatlimab in subjects with advanced and/or metastatic melanoma. There will be two arms to test the variables of ML NK cell source. ML NK cells from an autologous source will be used for Arm 1, and ML NK cells from an allogeneic source will be used for Arm 2. The investigators hypothesize that ML NK cells from either an autologous source or allogeneic source are safe and tolerable in subjects with advanced and/or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed advanced or metastatic melanoma that has progressed after at least 12 weeks or a minimum of 2 doses of treatment with a standard of care PD1/PDL1 containing therapy (nivolumab, pembrolizumab, atezolizumab, or durvalumab).
* Age: ≥18 years of age
* Have an Eastern Cooperative Oncology Group Performance Status (ECOG) ≤ 2 at screening Form Arm 1 only: Patients must meet the eligibility criteria to undergo apheresis to obtain autlogous NK cells.
* For Arm 2 only: Patient must have an available allogeneic NK cell donor who meets the eligibility criteria.
* Adequate organ function as defined below:

  * Total bilirubin < 2 mg/dL
  * AST(SGOT)/ALT(SGPT) < 3.0 x ULN
  * Creatinine within normal institutional limits OR creatinine clearance > 40 mL/min/1.73 m^2 by Cockcroft-Gault Formula
  * Oxygen saturation ≥ 90% on room air
  * Ejection fraction ≥ 45%
* Patients with a prior history of symptomatic CNS metastases must have received treatment and be neurologically stable for at least for 4 weeks and off anti-seizure medication and steroids for 7 days prior to initiation of LDC.
* Able to be off corticosteroids and any other immune suppressive medications for at least 14 days prior to apheresis or lymphodepletion and continuing until 30 days after the infusion of the ML NK cells. However, use of physiological dosing of corticosteroids (defined as ≤15mg prednisone or equivalent) is permitted if deemed medically necessary.
* Women of childbearing potential must have a negative pregnancy test within 28 days prior to study registration. Female and male patients (along with their female partners) must agree to use two forms of acceptable contraception, including one barrier method, throughout participation in the study and for at least 5 months after the last dose of relatlimab.
* Life expectancy >12 weeks
* Ability to understand and willingness to sign an IRB approved written informed consent document

Exclusion Criteria:

* Active autoimmune disorder requiring immunosuppression (physiologic steroids defined as ≤15mg prednisone or equivalent are acceptable).
* Prior history of an immune-related Grade 3 or 4 AE attributed to prior cancer immunotherapy (other than endocrinopathy managed with either replacement therapy or asymptomatic elevation of serum amylase or lipase) that resulted in permanent discontinuation of the prior immunotherapeutic agent.
* Patients with Grade ≤2 irAE who have not completely recovered from irAE (i.e. have residual toxicities >Grade 1) related to prior cancer immunotherapy (other than endocrinopathy management with replacement therapy or stable vitiligo). Patients treated with corticosteroids for irAE must demonstrate absence of related signs or symptoms for ≥7 days following discontinuation of corticosteroids.
* Leptomeningeal disease, carcinomatous meningitis, or symptomatic CNS metastases. Patients with asymptomatic brain metastasis with no pending intervention needed, or patients with treated CNS disease and stable for at least 4 weeks and off anti-seizure medication and steroids for 7 days prior to initiation of LDC are eligible.
* Known hypersensitivity to one or more of the study agents.
* Comorbidities and any conditions, that in the opinion of the investigator, that put the subject at unacceptable risk for study therapy or prevent the participant from consenting or participating in the study.
* Uncontrolled and active systemic infections, including but not limited to HIV, Hepatitis B or C infection.
* Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
* New progressive pulmonary infiltrates concerning for new or uncontrolled infectious process. Infiltrates attributed to infection must be stable/ improving after 1 week of appropriate therapy (4 weeks for presumed or proven fungal infections).
* Received any investigational or off-label drugs, or cytotoxic chemotherapy within the 14 days or five half-lives (whichever is greater) prior to apheresis.
* Pregnant or breastfeeding.
* Subjects are not acceptable candidates if they received prior tumor infiltrating lymphocytes (TIL) therapy (either in the setting of clinical trial or standard of care if TIL therapy is FDA approved in the future), or an organ allograft.
* Has a known additional malignancy that is progressing or required active treatment within the past 2 years. Note: participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg. Breast carcinoma, cervical cancer in situ) that has undergone potentially curative therapy are not excluded.
* Received a live or attenuated vaccine within 28 days prior to the beginning of the lymphodepletion therapy.

Eligibility Criteria for Haploidentical Donors (For Arm 2 only)

* Donor must be at least 18 years of age.
* Donor must be willing, in general good health, and medically able to tolerate leukapheresis required for harvesting the NK cells for this study.
* Donor must be negative for hepatitis, HTLV, and HIV on donor viral screen.
* Donor may not be pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 30 days prior to apheresis.
* Donor must be able to understand and willing to sign an IRB-approved written informed consent document.
* Only haploidentical donors will be included.
* Donor must meet the requirements of institutional donor guidelines, including the requirements of Foundation for the Accreditation of Hematopoietic Cell Therapy (FACT) criteria.

Eligibility Criteria for Autologous Patients (For Arm 1 only)

* Patient must be willing and medically able to tolerate leukapheresis required for harvesting the NK cells for this study.
* Patient must be negative for hepatitis, HTLV, and HIV on the viral screen.
* Patient may not be treated with any cytotoxic treatment within 2 weeks prior to leukapheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
For treatment with cells from an autologous source: Incidence and severity of adverse events | From start of treatment through end of safety follow-up (estimated to be 15 months)
  -As determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
For treatment with cells from an allogeneic source: Incidence and severity of adverse events | From start of treatment through end of safety follow-up (estimated to be 15 months)
  -As determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through completion of treatment (estimated to be 12 months)
  Objective response rate (ORR), defined as the proportion of patients with a complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, according to RECIST v1.1. 4 weeks apart.
  * Complete Response (CR). Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm).Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR). At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Duration of response (DOR) | Through completion of follow-up (estimated to be 3 years)
  -Duration of response (DoR), defined as the time from the first occurrence of a documented response after the ML NK cell infusion, to disease progression according to RECIST v1.1 or death.
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 3 years)
  * PFS, defined as the time from ML NK cell infusion to the first occurrence of disease progression according to RECIST 1.1 or death from any cause.
  * Progressive Disease (PD). At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm). Appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Disease control rate (DCR) | Through completion of follow-up (estimated to be 3 years)
  * Disease control rate (DCR), defined as the percentage of patients who have achieved a complete response, partial response, or stable disease according to RECIST v1.1.
  * Complete Response (CR). Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm).Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR). At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD). Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Overall survival (OS) | Through completion of follow-up (estimated to be 3 years)
  -OS, defined as the time from ML NK cell infusion to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Y Zhou, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu